CLINICAL TRIAL: NCT05329831
Title: Determining the Effect of Telehealth Education Intervention Given to Lupus Patients on Pain, Happiness and Life Activities: A Randomized Controlled Study
Brief Title: Effects of Telehealth Initiative on Lupus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Halil Ibrahim Tuna PhD, Principal Investigator, Selcuk University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LUPUS-1
Record Dates: First submitted 2022-02-03; First posted 2022-04-15 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Life activities; Pain; Happiness
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Pain

STUDY DESIGN:
Intervention Model Description: randomized controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Patients will be asked to fill out the Introductory Information Form, the Numerical Rating Scale, the Oxford Happiness Scale Short Form, and the Life Activities Scale scales. Then, the educational needs of the patients in the experimental group will be determined. Trainings will be planned individually for each patient according to the needs of the patients.
  After the patients go to their homes, telehealth will be implemented. Patients included in the experimental group will continue their routine physician appointments and prescriptions. In addition, telehealth education initiative will be made for the patients. Structured training will be applied to the patients once a week for 12 weeks, each training will be 20-40 minutes. The researcher will develop a trusting relationship with the patient and evaluate the patient's compliance with treatment, obstacles to happiness, information needs related to pain management, and difficulties in life activities.
  Interventions: Behavioral: Structured training using telehealth
- Control (No Intervention): No application will be made by the researcher to the patients in the control group. Patients will continue with their prescriptions and physician visit routines. The scales will be administered to the patients in this group at the beginning of the study and at the 4th, 8th, and 12th weeks.

INTERVENTIONS:
Behavioral: Structured training using telehealth — The intervention is based on self-care activities. Self-care states that people have an innate ability to take care of themselves.
  Arms: Experimental

SUMMARY:
SLE is mostly seen in young women and causes significant deformity in patients. In SLE, disease activity, body damage due to disease or treatment, comorbidities, and drugs affect body image negatively. SLE causes changes in the body such as skin rashes, uneven pigmentation, vitiligo, scars, tooth loss, alopecia, increased facial hair, stretch marks, weight gain, fatigue, pain, depression, the unpredictability of exacerbations or lack of independence, which worsens the subjective well-being of patients. can affect in that direction. Subjective well-being (SBL) is the scientific term for happiness, and SLE is thought to have a significant negative impact on SWB.

DETAILED DESCRIPTION:
Telehealth has been proposed as a component of patient education for disease management. Telehealth, which is defined as the remote delivery of health services via telecommunication tools including telephone and internet, enables accessible and appropriate health care service and provides communication, support, and monitoring opportunities with patients. Researchers think that a telehealth education initiative can be effective on the pain and life activities of SLE patients and this effect will improve their happiness in a good way. Based on these findings, this study aimed to examine the effects of a specific telephone educational intervention on pain, happiness, and activities of living in patients with SLE. The hypothesis of this study is; is that adapted telehealth education intervention can increase the happiness and life activities of patients with SLE and reduce pain.

ELIGIBILITY:
Inclusion Criteria:

* Those between the ages of 18-45,
* Diagnosed with SLE disease
* Those who are in remission of the disease
* Those who do not use biological DMARDs
* Non-smokers
* Those who do not drink alcohol
* Those with low disease activity score,
* Neurological, psychiatric disease and non-malignant,
* Individuals who are literate, able to communicate verbally and agree to participate in the study, among those evaluated and approved by their physicians.

Exclusion Criteria:

* Having a chronic disease other than SLE
* Having a rheumatological disease other than SLE
* Having a disability to use the phone
* Those with hearing loss or visual impairment,
* Those who have undergone changes in the treatment process and those who practice non-drug therapy during the study will not be included in the study.

In determining the inclusion, exclusion and termination criteria, both the literature and the consultation of a specialist in the field were taken.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale | 12 weeks
  It is a form that includes numbers and is used in grading pain. The intensity of pain felt by the patient is marked on a 10 cm ruler, with painlessness (0: no pain) at one end and the most severe pain possible (10: most severe pain) at the other end.

SECONDARY OUTCOMES:
Life Activity Scale | 12 weeks
  The index identifies activities aimed at providing the basic requirements necessary for the maintenance of life. The ADL index consists of a total of six questions containing information about bathing, dressing, toilet, movement, excretion and feeding activities. The individual is evaluated by giving 3 points if he/she does the activities of daily living independently, 2 points if he/she does it with help, and 1 point if he/she cannot do it at all. In the ADL index, 0-6 points are evaluated as dependent, 7-12 points as "semi-dependent", and 13-18 points as "independent".
Oxford Happiness Scale Short Form | 12 weeks
  The scale is a 7-item 5-point Likert type (1-Strongly Disagree, 5-Totally Agree) self-report scale. The highest score that can be obtained on the scale is 35, and the lowest score is 7. A high score indicates that subjective well-being is high.

CONTACTS AND LOCATIONS:
Locations (1):
- Selcuk University Hospital, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It may be considered later in the research.